CLINICAL TRIAL: NCT05329428
Title: PREDIN: Pregnancy and Vitamin D Intervention Study - A Randomized Controlled Trial
Brief Title: PREDIN: Pregnancy and Vitamin D Intervention Study
Acronym: PREDIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-03871
Record Dates: First submitted 2021-12-09; First posted 2022-04-15 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Vitamin D Deficiency; Vitamin D3 Deficiency; Pregnancy Complications
MeSH Terms: conditions — Vitamin D Deficiency; Pregnancy Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vitamin D Supplementation 20 µg/day (Experimental): Dietary supplements containing 20 µg of vitamin D per day will be provided to study subjects.
  Interventions: Dietary Supplement: Vitamin D Supplementation 20 µg/day
- Vitamin D Supplementation 40 µg/day (Experimental): Dietary supplements containing 40 µg of vitamin D per day will be provided to study subjects.
  Interventions: Dietary Supplement: Vitamin D Supplementation 40 µg/day
- Usual Antenatal Care (Active Comparator): Women randomized to usual antenatal care will receive advise about vitamin D supplementation according to usual antenatal care routines.
  Interventions: Other: Usual Antenatal Care

INTERVENTIONS:
Dietary Supplement: Vitamin D Supplementation 20 µg/day — At a routine visit at the antenatal care in early pregnancy (gestational week <15) women will be provided with with vitamin D3 (cholecalciferol) supplements. Two tablets, with a total content of 20 µg (800 IE), are taken daily throughout pregnancy.
  Arms: Vitamin D Supplementation 20 µg/day
Dietary Supplement: Vitamin D Supplementation 40 µg/day — At a routine visit at the antenatal care in early pregnancy (gestational week <15) women will be provided with with vitamin D3 (cholecalciferol) supplements. Two tablets, with a total content of 40 µg (1600 IE), are taken daily throughout pregnancy.
  Arms: Vitamin D Supplementation 40 µg/day
Other: Usual Antenatal Care — In early pregnancy (gestational week <15) women are advised by the regular midwife to take a daily supplement of Vitamin D throughout pregnancy, according to usual antenatal care routines.
  Arms: Usual Antenatal Care

SUMMARY:
Vitamin D deficiency is common among certain risk groups in Sweden, and occurs approximately in every tenth pregnant woman.The aim of the randomized double-blind controlled trial Pregnancy vitamin D intervention (PREDIN) is to investigate the dose of vitamin D supplementation required in achieving vitamin D sufficiency (25OHD ≥50 nmol/l) in pregnant women at risk of vitamin D deficiency. In addition, the investigators aim to examine if the overall vitamin D status and vitamin D intake have increased since the expanded vitamin D fortification program was initiated in year 2020.

DETAILED DESCRIPTION:
The effect of maternal vitamin D in pregnancy for maternal and offspring health needs to be clarified. In observational studies, the investigators and others show associations between poor maternal vitamin D status in pregnancy and an increased risk of pregnancy complications. Poor maternal vitamin D status is also linked to impaired growth in the first year of life, and potentially also to higher risk of developing obesity in childhood. Risk factors for vitamin D deficiency in Swedish pregnant women are related to lower intake of vitamin D and to less sun exposure.

Since the evidence for positive effects of maternal vitamin D status or intake is limited, vitamin D interventions in pregnancy are warranted to clarify the causal effects of vitamin D in pregnancy and the doses required to achieve sufficient vitamin D status in deficient women. In the first trimester, pregnant women will be screened at a routine visit in the antenatal care for the risk of vitamin D deficiency using a validated questionnaire. Women who are classified as having a high risk of vitamin D deficiency will be randomized to one of three study arms: usual antenatal care, 20 µg vitamin D per day or 40 µg vitamin D per day. The participants will be followed up until delivery. Blood will be collected for analysis of vitamin D status (25OHD) at screening and in the third trimester of pregnancy. Information regarding pregnancy, gestational complication and fetal growth will be retrieved from medical records after delivery. About 500 women will be screened and their vitamin D status and vitamin D intake will be compared to a previous population-based cohort study, to investigate if the status or intake of vitamin D has increased since the expanded food fortification program was introduced.

The study hypothesis is that vitamin D status and/or vitamin D intake is related to risk of developing complications during pregnancy or delivery and that maternal supplementation with vitamin D during pregnancy will be effective in achieving vitamin D sufficiency in pregnant women at risk of vitamin D deficiency. In addition, the investigators hypothesize that the expanded vitamin D food fortification program has increased the vitamin D status and vitamin D intake of pregnant women in Gothenburg since 2013-2014.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women in gestational week <15

Exclusion Criteria:

* multi-fetal pregnancy
* known disorder to the metabolism of vitamin D, calcium or phosphate (e.g. adrenal gland disorders, kidney disease)
* ongoing treatment with vitamin D of ≥10 µg/day
* difficulties understanding the study information

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Difference in maternal vitamin D status (25OHD) between intake of vitamin D supplements containing either 40 µg per day or 20 µg per day during pregnancy | From inclusion in first trimester to follow-up in third trimester, up to 9 months
  Analyses of 25OHD (25OHD3 and 25OHD2) from blood samples drawn in first- and third trimester of pregnancy
Difference in maternal vitamin D status (25OHD) between intake of vitamin D supplements (both 40 µg per day or 20 µg per day) during pregnancy and usual antenatal care routines | From inclusion in first trimester to follow-up in third trimester, up to 9 months
  Analyses of 25OHD (25OHD3 and 25OHD2) from blood samples drawn in first- and third trimester of pregnancy
Difference in maternal 3-epi-25-Hydroxyvitamin D between the three groups; intakes of vitamin D supplements 40 µg/day or 20 µg/day or usual antenatal care routines | From inclusion in first trimester to follow-up in third trimester, up to 9 months
  Analyses of vitamin D metabolites 3-epi-25-Hydroxyvitamin D3 from blood samples drawn in first- and third trimester of pregnancy
Difference in maternal 1,25-dihydroxyvitamin D between the three groups; intakes of vitamin D supplements 40 µg/day or 20 µg/day or usual antenatal care routines | From inclusion in first trimester to follow-up in third trimester, up to 9 months
  Analyses of 1,25-dihydroxyvitamin D from blood samples drawn in first- and third trimester of pregnancy
Difference in maternal vitamin D binding proteins between the three groups; intakes of vitamin D supplements 40 µg/day or 20 µg/day or usual antenatal care routines | From inclusion in first trimester to follow-up in third trimester, up to 9 months
  Analyses of vitamin D binding proteins from blood samples drawn in first- and third trimester of pregnancy

SECONDARY OUTCOMES:
Gene variant related to vitamin D metabolism | At inclusion in first trimester of pregnancy
  Analyses of gene variants in blood sample drawn at inclusion in first trimester of pregnancy
Ferritin | From inclusion in first trimester to follow-up in third trimester, up to 9 months
  Analyses of ferritin
Hemoglobin | From inclusion in first trimester to follow-up in third trimester, up to 9 months
  Analyses of hemoglobin
Metabolomics | From inclusion in first trimester to follow-up in third trimester, up to 9 months
  Analyses of metabolomics in blood
C-reactive protein | From inclusion in first trimester to follow-up in third trimester, up to 9 months
  Analyses of inflammation e.g. c-reactive protein
Interleukines | From inclusion in first trimester to follow-up in third trimester, up to 9 months
  Analyses of inflammation e.g. interleukines
Cytokines | From inclusion in first trimester to follow-up in third trimester, up to 9 months
  Analyses of inflammation e.g. cytokines
Cortisol | From inclusion in first trimester to follow-up in third trimester, up to 9 months
  Analyses of cortisol
Parathyroid hormone | From inclusion in first trimester to follow-up in third trimester, up to 9 months
  Analysis of parathyroid hormone in sampled blood at the routine laboratory
Estrogen | From inclusion in first trimester to follow-up in third trimester, up to 9 months
  Analyses of estrogen, in sampled blood, at the routine laboratory
Progesterone | From inclusion in first trimester to follow-up in third trimester, up to 9 months
  Analyses of progesterone, in sampled blood, at the routine laboratory
24,25-Dihydroxyvitamin D | From inclusion in first trimester to follow-up in third trimester, up to 9 months
  Analyses of 24,25(OH)2D (24,25(OH)2D3 and 24,25(OH)2D2)
Dietary intake | At inclusion in first trimester and at follow-up in third trimester, up to 9 months
  Dietary intake of mother during pregnancy assessed by dietary record at two time points
Body weight development | From inclusion in first trimester to follow-up in third trimester, up to 9 months
  Self-reported weight (in kilograms) during pregnancy until delivery.
Incidence of pregnancy-induced hypertension | Up to delivery
  Diagnosis of pregnancy-induced hypertension
Incidence of pre-eclampsia | Up to delivery
  Diagnosis of pre-eclampsia
Incidence of gestational diabetes | Up to delivery (up to 9 months)
  Diagnosis of gestational diabetes
Incidence of preterm delivery | Up to 37 completed weeks
  Delivery before 37 weeks completed weeks of gestation
Incidence of small for gestational age (SGA) | At delivery
  SGA born infant
Incidence of large for gestational age (LGA) | At delivery
  LGA born infant
Incidence of Intrauterine growth restriction (IUGR) | At delivery
  IUGR
Apgar scores | At 1, 5 and 10 minutes after delivery
  Vitality signs are estimated as Apgar scores at 1, 5 and 10 minutes after birth of the newborn. Apgar stands for Appearance, pulse, grimace, activity and respiration. The maximium score at each time point is 10 scores and a high score indicates high vitality, where as a low score indicates very low vitality.
Incidence of Caesarean sections | At delivery
  Delivery by caesarean sections
Incidence of miscarriage | During the first 21+6 weeks of pregnancy
  Miscarriage
Incidence of Intrauterine fetal demise (IUFD) | Any time during pregnancy after pregnancy week 22+0 (up to 9 months)
  IUFD

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Augustin, Ass Prof, Principal Investigator — Göteborg University
Locations (1):
- Antenatal Care, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT05329428/Prot_SAP_000.pdf